CLINICAL TRIAL: NCT01068067
Title: Validation of Pharmacogenetics Plus Drug Combination Guided Initial Tacrolimus Dosage in Chinese Renal Transplant Recipients: A Prospective Randomized Controlled Study
Brief Title: Validation of Pharmacogenetics Plus Drug Combination Guided Initial Tacrolimus Dosage in Renal Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Min Huang, School of Pharmaceutical Sciences, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAC+WUZHI
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-01

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Pharmaceutical Preparations; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pharmacogenetics plus SchE guided dosing (Experimental)
  Interventions: Other: drug (tacrolimus and SchE) and genetics
- standard dosing (Active Comparator)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Other: drug (tacrolimus and SchE) and genetics — Patients were genotyped for the polymorphisms that can influence tacrolimus pharmacokinetics before transplantation. After transplantation, initial tacrolimus dosage was based on an algorism guided by pharmacogenetics and SchE.
  Arms: pharmacogenetics plus SchE guided dosing
Drug: tacrolimus — After transplantation, patients received standard initial dose of tacrolimus (0.050-0.075 mg/kg).
  Arms: standard dosing

SUMMARY:
The purpose of this study is to compare pharmacogenetics plus drug combination (Schisandra sphenanthera extract,SchE)guided and standard initial tacrolimus dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (both males and females, 18-65 years) recipients underwent single primary renal transplantation in the First Affiliated Hospital of Sun Yat-sen University
2. Wish to participate in the study
3. Informed consent for the trial

Exclusion Criteria:

1. Patients with abnormal hepatic function, serious infection, malignant tumour, and diabetes mellitus
2. Patients with ABO-incompatible renal transplantation
3. Panel reactive antibody (PRA) levels greater than 30% before transplantation
4. Underwent combined organ transplantations
5. Except for SchE, other medication known to affect tacrolimus blood levels, such as diltiazem, verapamil, ketoconazole, itraconazole, erythromycin or clarithromycin was used
6. Allergic history to study medicines
7. During pregnancy or plan to get pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
C0 of tacrolimus after the initial dose, the percentage of out-of-range C0 after initial dose, the number of dose adjustments made to achieve therapeutic range (5-10 ng/ml) and the dose requirement to reach therapeutic range | not less than three days after initial dose and not more than one month

SECONDARY OUTCOMES:
acute rejection rate within two weeks after transplantation | within two weeks after transplantation
serum creatinine at fourteen days after transplantation | fourteen days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Min Huang, PhD, Study Chair — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University; Chang-Xi Wang, MD, Study Director — Kidney Transplant Department, Transplant Center, the First Affiliated Hospital of Sun Yat-sen University; Jia-Li Li, PhD, Principal Investigator — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University; Xue-Ding Wang, MD, Principal Investigator — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University; Si-Yang Chen, MM, Principal Investigator — Anesthesia Department, the First Affiliated Hospital of Sun Yat-sen University
Locations (2):
- China (2):
  - Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, Guangdong
  - Kidney Transplant Department, Transplant Center, the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong

REFERENCES:
- See also: Help Me Understand Genetics — http://ghr.nlm.nih.gov/handbook
- See also: Cytochrome P450 — http://ghr.nlm.nih.gov/glossary=cytochromep450
- See also: Tacrolimus — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a601117.html
- See also: Kidney (Renal) transplantation — http://en.wikipedia.org/wiki/Kidney_transplantation